CLINICAL TRIAL: NCT06649058
Title: EXCLAIM: Exploring Combined Local and Systemic Approaches In Brain Metastasis: a Multi-cohort Randomized Phase II Study Evaluating Initial Response to Systemic Therapy and Subsequent Integration of Stereotactic Radiosurgery in Patients With Low-risk Brain Metastases and Central Nervous System-active Systemic Therapy Options
Brief Title: EXCLAIM: Exploring Combined Local and Systemic Approaches In Brain Metastasis: a Multi-cohort Randomized Phase II Study Evaluating Initial Response to Systemic Therapy and Subsequent Integration of Stereotactic Radiosurgery in Patients With Low-risk Brain Metastases and Central Nervous System-active
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1383; NCI-2024-08780 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- cSRS PR or SD (Experimental): Patients with a CR will be observed with ongoing standard of care MRI. Patients with SD or PR will be randomized to receive cSRS or ongoing observation.
  Interventions: Other: Systemic Therapy; Radiation: Stereotactic Radiosurgery
- a-pdSR CNS PD (Experimental): At the time of CNS PD, patients will also be randomized to pdSRS versus pdSRS + cSRS.
  Interventions: Other: Systemic Therapy; Radiation: Stereotactic Radiosurgery
- b-PDC CNS PD (Experimental): At the time of CNS PD, patients will also be randomized to pdSRS versus pdSRS + cSRS.
  Interventions: Other: Systemic Therapy; Radiation: Stereotactic Radiosurgery
- SST treated SD or PR patients to receive cSRS/ ongoing observation (Experimental): Patients with a CR will be observed with ongoing standard of care MRI. Patients with SD or PR will be randomized to receive cSRS or ongoing observation.
  Interventions: Other: Systemic Therapy; Radiation: Stereotactic Radiosurgery
- SST treated PD patients to pdSRS / pdSRS+cSRS (Experimental): At the time of CNS PD, patients will also be randomized to pdSRS versus pdSRS + cSRS.
  Interventions: Other: Systemic Therapy; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Other: Systemic Therapy — Participants will receive systemic therapy as a standard of care therapeutic option
Radiation: Stereotactic Radiosurgery — Participants will receive systemic therapy as a standard of care therapeutic option

SUMMARY:
To learn if consolidative stereotactic radiosurgery (cSRS) can help to control central nervous system (CNS) disease in patients who have brain metastases and have a partial response or stable brain metastases after systemic therapy.

To learn if using SRS to treat all brain metastases that do not respond to systemic therapy versus treating only metastases that are getting worse can help to control CNS disease in patients whose disease gets worse after systemic therapy.

DETAILED DESCRIPTION:
Primary Objectives:

To assess whether cSRS improves CNS progression-free survival (CNS-PFS) in patients with BM who have a PR or SD with upfront systemic therapy.

To assess whether SRS to all BM not in CR (cSRS + pdSRS) versus only progressing lesions (pdSRS) improves CNS-PFS in patients with CNS progression on upfront systemic therapy.

Secondary Objectives:

To report the rate and degree of response of BM to systemic therapy by specific regimen and histology.

To report adverse neurologic events that occur with BM treated with upfront systemic therapy and differences in these events between various downstream radiation therapy options (omission, cSRS, pdSRS, etc).

To evaluate rates of LMD in all patients managed with upfront systemic therapy and differences in LMD rates between various downstream radiation therapy options (omission, cSRS, pdSRS, etc).

To evaluate neurocognitive changes in patients treated with upfront systemic therapy for BMand differences in these changes between various downstream radiation therapy options (omission, cSRS, pdSRS, etc).

To perform inference on overall survival as estimated by the Kaplan-Meier estimator in patients treated with upfront systemic therapy for BM and differences in these changes between various downstream radiation therapy options (omission, cSRS, pdSRS, etc).

Exploratory Objectives:

To correlate imaging biomarkers with outcomes of BM treated with systemic therapy.

To correlate volumetric assessment of lesion response to conventional assessment by mRECIST 1.1.

To explore ML as a tool to predict outcomes of BM treatment based on disease specific, clinical, and lesion specific features.

To explore the association of circulating bioanalytes with up front systemic therapy for BM and subsequent downstream management strategies (i.e. cSRS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Evaluation by a brain metastasis multidisciplinary team (BM-MDT) consisting of a medical oncologist (can be the patient's primary medical oncologist), a radiation oncologist who regularly performs SRS, and a neurosurgeon. This evaluation can take place in clinic or during a multidisciplinary conference.
3. Life expectancy > 6 months as estimated by BM-MDT.
4. BM-MDT agreement that the planned systemic therapy regimen may provide intracranial benefit (SD, PR, or CR in the CNS).
5. BM-MDT agreement that the patient's BM does not require immediate local therapy (surgery and/or radiation therapy); i.e. it is judged to be safe to omit local therapy as initial BM management.
6. The patient's BM are amenable to SRS as initial local therapy as determined by BM-MDT.
7. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
8. Histologically confirmed metastatic cancer with at least one measurable metastasis in the brain (≥ 5 mm).
9. At least one measurable intracranial target lesion which was not previously treated with SRS. Regrowth in a cavity of previously excised lesion will not qualify as a measurable lesion. Growth or change in a lesion previously irradiated will not qualify as a measurable lesion.
10. Prior SRS and prior excision of BM is permitted if other measurable non irradiated lesions as described in #9 remain.
11. The resection cavity of excised BM must have received appropriate radiation therapy (pre or post operative SRS, brachytherapy) or have been observed for >6 months after resection without evidence of local cavity recurrence.
12. Subjects must be free of neurologic signs and symptoms related to metastatic brain lesions either without systemic corticosteroids or requiring ≤ 2 mg dexamethasone daily for symptom resolution.
13. ECOG performance status ≤ 1.
14. Documented agreement by the patient's primary medical oncologist with the appropriateness of planned SST regimen.
15. This study will allow non-English speaking subjects to be enrolled. Verbal Translation Preparative Sheet (VTPS) will be used if a translated consent form is not available in the subject's language. The consent form will be translated into the language of the subject after 2 or more occurrences. This will apply to any MD Anderson patient.

Exclusion Criteria:

1. History of known leptomeningeal involvement (radiographic or cytological).
2. Small cell lung cancer, lymphoma, or leukemia histology.
3. Non-small cell lung cancer histology with targetable oncogenic driver mutation with planned initiation of highly CNS active targeted therapy (eg osimertinib, brigatinib, alectinib, or lorlatinib).
4. Subjects previously treated with WBRT.
5. Any intact BM size > 3 cm. After surgical excision and appropriate radiation therapy to the cavity, patients may enroll if additional eligible lesions are present.
6. Prior disease progression on one or more of the agents comprising SST.
7. Exposure to one or more agents comprising SST within the last 30 days.
8. Prior unacceptable toxicity during treatment with one or more agents comprising SST.
9. Subjects with a major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled.
10. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Note: The time requirement does not apply to participants who underwent successful treatment of superficial bladder cancer, in situ cervical cancer, ductal carcinoma in situ, or other in-situ cancers. Subjects with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
11. Skin Cancer Exclusion: Please note that localized cutaneous basal cell carcinoma and squamous cell carcinoma is not an exclusion criterion regardless of treatment status. Biopsy proven metastatic disease from these histologies is an exclusion criterion if this constitutes a second cancer.
12. Patient weight >450 pounds.
13. Patient had prior SRS to any intracranial lesion <15mm from a metastasis on the screening MRI. Prior MRIs and DICOMs will be used to make this determination.
14. Patient unable to receive a brain MRI (implanted metal devices or foreign bodies) or MRI contrast.
15. Any BM with a significant hemorrhagic component (defined as MRI T1 intrinsic hyperintensity comprising ≥ 25% of maximal lesion diameter).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Beckham, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org